CLINICAL TRIAL: NCT04247646
Title: SLeep and OPioid UsE in Patients Undergoing Total Knee Arthroplasty
Acronym: SLOPE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Scripps Health (Other)
Responsible Party: Principal Investigator, Stuti Jaiswal, Faculty Hospitalist, Scripps Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 65106563709047
Record Dates: First submitted 2020-01-27; First posted 2020-01-30 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Opioid Use; Pain, Postoperative; Sleep; Delirium
MeSH Terms: conditions — Pain, Postoperative; Delirium | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Melatonin (Active Comparator): Melatonin 5 mg sublingual nightly x 29 nights, starting on post-operative day 0.
  Interventions: Dietary Supplement: Melatonin
- Placebo (Placebo Comparator): Placebo troche, sublingual nightly x 29 nights, starting on post-operative day 0.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Melatonin — Participants will take sublingual melatonin (or placebo) nightly for 29 doses after undergoing total knee replacement surgery.
  Arms: Melatonin
Dietary Supplement: Placebo — Participants will take sublingual melatonin (or placebo) nightly for 29 doses after undergoing total knee replacement surgery.
  Arms: Placebo

SUMMARY:
Prescription opioid misuse and its associated negative effects have become an epidemic in the United States, and post-operative opioid use contributes to this terrible problem. Alternative strategies to opioid prescribing are thus highly sought after in the post-operative setting. Importantly, sleep and pain have a bi-directional relationship, and inadequate or impaired sleep regularly occur following orthopedic operations. Melatonin is an endogenous sleep hormone that can be administered exogenously, and that has been shown to have some potential as an analgesic agent. Here, using the premise that melatonin may improve sleep and pain in the post-operative setting, the investigators propose a randomized clinical trial in 120 participants undergoing total knee arthroplasties. Patients will be randomized to receive either sublingual melatonin 5 mg or matched placebo starting on post-operative day (POD) 0 and through POD . The investigators will measure post-operative opioid usage as the primary outcome, and post-operative pain scores as a secondary outcome. The primary safety outcome will be sedation level, as measured by the Richmond Agitation Sedation Scale (RASS). Sleep will be measured objectively using wrist-worn actigraphy. Participants will be followed through POD 28, and will also have baseline data on sleep, pain, and cognition obtained prior to surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 years and older
* Undergoing elective total knee arthroplasty (single knee)

Exclusion Criteria:

* Non-English speakers
* Individuals with dementia
* Patients with liver cirrhosis
* Patients currently taking prescription sleep aids
* Patients with long-term (greater than 3 months prior to surgery), chronic opioid use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Opioid use | Post-operative day 0 through post-operative day 28
  morphine milligram equivalents of opioid medications used by the participant

SECONDARY OUTCOMES:
Pain level | Post-operative day 0 through post-operative day 28
  Numerical pain scores reported by the patient following surgery using the Visual Analog Scale (Scale of 0-10, with 0 being no pain and 10 being the worst possible pain).
Other pain medicine usage | Post-operative day 0 through post-operative day 28
  Usage of non-opioid analgesics used by the participant
Total daily sleep duration | Post-operative day 0 through post-operative day 28
  Minutes of sleep obtained daily as measured by actigraphy
Nightly sleep duration | Post-operative day 0 through post-operative day 28
  Minutes of sleep obtained nightly as measured by actigraphy
Sleep fragmentation | Post-operative day 0 through post-operative day 28
  Mean/median length of the sleep bout during nightly sleep

OTHER OUTCOMES:
Delirium Incidence | Post-operative day 0 through hospital discharge
  Rates of inpatient delirium as measured by the Confusion Assessment Method
Change in sleep duration pre and post-operatively | Post-operative day 0 through post-operative day 28
  change in sleep duration (minutes) following surgery, using pre-operative sleep data as the comparator
Sedation levels | Post-operative day 0 through post-operative day 28
  Sedation levels, as measured by the Richmond Agitation Sedation Scale (RASS), during inpatient stay. RASS scores are measured on a scale of -5 to +5 with -5 equating to deeply sedated (deep coma) and +5 equating to extremely agitated/combative.
Subjective sleep | Post-operative day 0 through post-operative day 28
  subjective sleep scores as measured by the Richards Campbell Sleep Questionnaire while inpatient. The Richards Campbell Sleep Questionnaire is a 5-item questionnaire scored on a visual, 100 milimeter scale where the participants marks or selects where they fell on the scale in response to the specific question. Scores are assigned from 0-100 based on where the participant's response lies, with a higher score indicating better sleep.
Delirium incidence in those with elevated obstructive sleep apnea risk | Post-operative day 0 through post-operative day 28
  Delirium incidence in those with elevated OSA risk, based on the Berlin and STOP-BANG criteria

CONTACTS AND LOCATIONS:
Overall Officials: Stuti Jaiswal, MD PhD, Principal Investigator — Scripps Clinic Medical Group
Locations (1):
- Scripps Green Hospital, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Undecided